CLINICAL TRIAL: NCT03323671
Title: Preemptive Analgesia for Primary Dysmenorrhoea: a Randomized Controlled Trial
Brief Title: Preemptive Analgesia for Primary Dysmenorrhoea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hanan Nabil (Other)
Responsible Party: Sponsor-Investigator, Hanan Nabil, Associate Professor Obstetrics and Gynecology, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 27011975
Record Dates: First submitted 2015-10-27; First posted 2017-10-27 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Primary Dysmenorrhea
Keywords: primary dysmenorrhea; preemptive analgesia
MeSH Terms: interventions — Mefenamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- premenstruation group (Experimental): preemptive mefenamic acid 500mg tablets every 8 hours starting 2 days before anticipated menstruation and during the first 2 days of the cycle
  Interventions: Drug: preemptive mefenamic acid
- menstruation group (Experimental): mefenamic acid 500mg tablets every 8 hours during the first 2 days of the cycle
  Interventions: Drug: mefenamic acid

INTERVENTIONS:
Drug: preemptive mefenamic acid — preemptive analgesia before menstrual pain
  Other Names: ponstan forte
  Arms: premenstruation group
Drug: mefenamic acid — mefenamic acid given only during menstruation
  Other Names: ponstan forte
  Arms: menstruation group

SUMMARY:
Preemptive analgesia before the release of pain mediators

DETAILED DESCRIPTION:
spasmodic dysmenorrhea is one of the most distressing symptoms in women. adolescents shows a usual absence from school . prostaglandin release is one of the most accepted theory responsible for spasmodic dysmenorrhea.

Non steroidal anti inflammatory Drugs were proved to be one of the alternative medications for spasmodic dysmenorrhea.

Getting the idea of what is called preemptive anesthesia by blocking the receptors before catching pain mediators the study participants will be divided randomly into 2 group group 1 receiving ttt 2 days before the anticipated menstruation and group 2 receiving ttt only during menstruation as analgesia

ELIGIBILITY:
Inclusion Criteria:

* nulliparous ladies
* with regular menstrual cycle pattern
* those experienced history of dysmenorrhea (primary or spasmodic)
* patients able to sallow tables

Exclusion Criteria:

* irregular cycles
* any associated local causes( pelvic infection, endometriosis, fibroid or others)
* patients with familial Mediterranean fever or other intermenstrual attacks of abdominal pain
* gastric or duodenal ulcers or gastritis
* other contraindications to non steroidal anti-inflammatory drugs
* patients with severe diminution of vision or color discrimination
* patients with any depressive or mood disorders
* patients receiving any hormonal treatment

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
change in the Degree of pain | 4 months
  severity of pain according to visual pain analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Nabil, MD, Principal Investigator — Manoura University Hospital
Locations (1):
- Mansoura University, Al Mansurah, Egypt